CLINICAL TRIAL: NCT00796510
Title: A Phase 3, Multi-Center, Open Label Study To Evaluate The Long-Term Safety Of Monotherapy Sitaxsentan Sodium And Combination Therapy With Sitaxsentan Sodium And Sildenafil Citrate In Subjects With Pulmonary Arterial Hypertension
Brief Title: Study Providing Monotherapy (Sitaxsentan) And Combination Therapy (Sitaxsentan+Sildenafil) To Subjects With Pulmonary Arterial Hypertension (PAH) To Assess Long-Term Safety
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Safety Issue: The trial was prematurely terminated on Dec 9, 2010, due to safety concerns, specifically new emerging evidence of hepatic injury
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1321002
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Results first posted 2012-02-20 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Hypertension
Keywords: endothelin receptor antagonist (ETRA); sitaxsentan
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — sitaxsentan; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitaxsentan (Experimental): Monotherapy arm
  Interventions: Drug: Sitaxsentan
- Sitaxsentan and Sildenafil (Experimental): Combination treatment
  Interventions: Drug: Sitaxsentan and Sildenafil

INTERVENTIONS:
Drug: Sitaxsentan — Sitaxsentan = 100 mg tablet administered orally, once daily
  Arms: Sitaxsentan
Drug: Sitaxsentan and Sildenafil — Sitaxsentan = 100 mg tablet administered orally, once daily plus Sildenafil = 20 mg tablet administered orally, three times a day
  Arms: Sitaxsentan and Sildenafil

SUMMARY:
As sitaxsentan is the agent most highly selective for ETA (Endothelin Type A (receptor)), and does not significantly impact sildenafil pharmacokinetics the combination of most promise for pulmonary arterial hypertension (PAH) therapy is these two oral drugs administered in combination.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in B1321001 for at least 4 weeks.
* Previously enrolled in B1321003, discontinued from the study.
* Completed the B1321003 study as planned.

Exclusion Criteria:

* Treated with an investigational drug (other than sitaxsentan or sildenafil in either B1321001 or B1321003) or device that has not received regulatory approval within the 30 days prior to Baseline/Day 1 or during the study.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Fountain Valley, California, United States
- Pfizer Investigational Site, Cluj-Napoca, Romania
- Pfizer Investigational Site, Kyiv, Ukraine

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were previously enrolled in B1321001 (NCT00795639) or B1321003 (NCT00796666) only where pre-specified entry criteria were met.
Groups:
- Sitaxsentan: Sitaxsentan 100 milligrams (mg) orally once a day
- Sitaxsentan and Sildenafil: Sitaxsentan 100 mg daily and sildenafil 20 mg orally three times a day
Period: Overall Study
Arm/Group | Sitaxsentan | Sitaxsentan and Sildenafil
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Death | 1 | 0
Not completed — Study Terminated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitaxsentan | Sitaxsentan and Sildenafil | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Continuous [Mean (Full Range); unit: years] | 42.3 [29 to 54] |  | 42.3 [29 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is the duration from first dose to death. For participants who are lost to follow-up, survival was censored at the last date of follow-up.
Time Frame: Baseline and every 12 weeks up to Week 18
Population: Due to the premature termination only 3 participants were recruited into this study. No analyses were performed.
Arm/Group | Sitaxsentan | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in 6 Minute Walk Distance at Weeks 12 and 24
Description: The walk distance was the total distance walked during the 6-minute test. Change is distance walked at week x minus distance walked at baseline.
Time Frame: Baseline, Weeks 12 up to Early Termination (ET) (up to Week 18)
Population: Due to the premature termination only 3 participants were recruited into this study. No analyses were performed.
Arm/Group | Sitaxsentan | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants in Each World Health Organization (WHO) Functional Class of Pulmonary Arterial Hypertension (PAH)
Description: The WHO functional classes of PAH range from Class 1 (no limitation in physical activity) to Class IV (can not perform a physical activity without any symptoms).
Time Frame: Baseline, Week 12 and ET (up to Week 18)
Population: Due to the premature termination only 3 participants were recruited into this study. No analyses were performed.
Arm/Group | Sitaxsentan | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sitaxsentan | Sitaxsentan and Sildenafil
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/0
Other Adverse Events (participants affected / at risk) | 1/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (N=3) | Sitaxsentan and Sildenafil (N=0)
Cardiac arrest (Cardiac disorders) | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (N=3) | Sitaxsentan and Sildenafil (N=0)
Non-cardiac chest pain (General disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the premature termination only 3 participants were recruited into this study. No summarization or analysis was done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.